CLINICAL TRIAL: NCT04626947
Title: Prevention of Recurrent Clostridium Difficile Infection (CDI) in Patients With Inflammatory Bowel Disease (IBD).
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: David Binion, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, David Binion, MD, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY19100301
Record Dates: First submitted 2020-09-29; First posted 2020-11-13 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease; C. Diff. Infections
Keywords: C.diff; C. difficile; IBD; UC; Bezlotoxumab; Recurrent C. diff
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease; Clostridium Infections | interventions — bezlotoxumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open label (Other): Single arm
  Interventions: Biological: Bezlotoxumab

INTERVENTIONS:
Biological: Bezlotoxumab — Bezlotoxumab infusion

SUMMARY:
The study will compare the effectiveness of Bezlotoxumab in individuals with active C. diff ( Clostridium difficile) infection who are diagnosed with Inflammatory Bowel Disease.

DETAILED DESCRIPTION:
Bezlotoxumab is administered during a course of antibiotic therapy. The dose is administered as one time treatment. Patients will receive 10 mg/kg IV over 60 minutes as a single dose via central line.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* active CDI receiving therapy
* diagnosis of IBD
* and history of CDI.

Exclusion Criteria:

* <18 years old
* no IBD
* no CDI
* history of colectomy
* history of preexisting congestive heart failure
* pregnant or nursing women
* TCP<50
* past cardiac history.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Binion, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who are part of the IBD Registry and have a defined IBD diagnosis and CDI will be approached to be consented for this study.
Pre-assignment Details: Randomly the study treatment will be offered to 50 patients.
Groups:
- Open Label Bezlotuxumab: Single arm Bezlotoxumab infusion
Period: Overall Study
Arm/Group | Open Label Bezlotuxumab
Started | 19
90 Days | 17
12 Months | 8
Completed | 5
Not Completed | 14
Not completed — Study terminated | 14

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Bezlotuxumab
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19
IBD Type [Number; unit: participants]
  Crohn's disease (CD) | 14
  Ulcerative Colitis (UC) | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrent C. Diff Infection at 90 Days
Description: Rates of recurrent C. Diff infection defined by a positive molecular test for C. Diff and clinical symptoms.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Bezlotuxumab
Number analyzed (Participants) | 17
Participants | 1

2. Primary Outcome: Number of Participants With Recurrent C. Diff Infection at 12 Months
Description: Rates of recurrent C. Diff infection defined by a positive molecular test for C. Diff and clinical symptoms.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Bezlotuxumab
Number analyzed (Participants) | 8
Participants | 1

3. Primary Outcome: Number of Participants With Recurrent C. Diff Infection at 24 Months
Description: Rates of recurrent C. Diff infection defined by a positive molecular test for C. Diff and clinical symptoms.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Bezlotuxumab
Number analyzed (Participants) | 5
Participants | 0

4. Secondary Outcome: Number of Participants With Positive Inflammatory Markers After Bezlotuxumab Infusion 90 Days
Description: Rates of abnormal inflammatory markers C- Reactive protein (CRP) and Erythrocyte sedimentation rate (ESR) after 90 days from receiving Bezlotuxumab.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Bezlotuxumab
Number analyzed (Participants) | 17
Participants
  CRP | 6
  ESR | 8

5. Secondary Outcome: Number of Participants With Positive Inflammatory Markers After Bezlotuxumab Infusion 12 Months
Description: Rates of abnormal inflammatory markers C- Reactive protein (CRP) and Erythrocyte sedimentation rate (ESR) after 12 months from receiving Bezlotuxumab
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Bezlotuxumab
Number analyzed (Participants) | 8
Participants
  CRP | 0
  ESR | 0

6. Secondary Outcome: Number of Participants With Positive Inflammatory Markers After Bezlotuxumab Infusion 24 Months
Description: Rates of abnormal inflammatory markers C- Reactive protein (CRP) and Erythrocyte sedimentation rate (ESR) after 24 months from receiving Bezlotuxumab
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Bezlotuxumab
Number analyzed (Participants) | 5
Participants
  CRP | 1
  ESR | 1

7. Secondary Outcome: Quality of Life and Disease Activity Scores of Participants at Study Baseline
Description: Quality of life and disease activity scores at baseline. Short Inflammatory Bowel disease questionnaire (SIBDQ) Scores range 0-70 Higher scores represent better disease related quality of life. Harvey Bradshaw Index (HBI) for CD patients and Ulcerative colitis disease activity (UCAI) for UC patients. Score ranging from 0 to 20. Patients with a score of 3 or less likely to be in remission.
Time Frame: Index visit
Population: 14 CD, 5 UC
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label Bezlotuxumab
Number analyzed (Participants) | 19
score on a scale
  SIBDQ | 40.8 (14.02)
  HBI: number analyzed (Participants) | 14
  HBI | 8.6 (5.2)
  UCAI: number analyzed (Participants) | 5
  UCAI | 6.2 (5.7)

8. Secondary Outcome: Quality of Life and Disease Activity Scores of Participants After Bezlotuxumab Infusion 90 Days
Description: as for outcome 7
Time Frame: 90 Days
Population: CD=12, UC=5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label Bezlotuxumab
Number analyzed (Participants) | 17
score on a scale
  SIBDQ | 40 (18.08)
  HBI: number analyzed (Participants) | 12
  HBI | 6.5 (6.1)
  UCAI: number analyzed (Participants) | 5
  UCAI | 2.6 (1.8)

9. Secondary Outcome: Quality of Life and Disease Activity Scores of Participants After Bezlotuxumab Infusion 12 Months
Description: as for outcome 7
Time Frame: 12 months
Population: CD=7, UC=1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label Bezlotuxumab
Number analyzed (Participants) | 8
score on a scale
  SIBDQ | 49.75 (18)
  HBI: number analyzed (Participants) | 7
  HBI | 7.5 (5.6)
  UCAI: number analyzed (Participants) | 1
  UCAI | 3 (0)

10. Secondary Outcome: Quality of Life and Disease Activity Scores of Participants After Bezlotuxumab Infusion 24 Months
Description: as for outcome 7
Time Frame: 24 months
Population: CD=4, UC=1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label Bezlotuxumab
Number analyzed (Participants) | 5
score on a scale
  SIBDQ | 61.8 (6)
  HBI: number analyzed (Participants) | 4
  HBI | 3.7 (2.6)
  UCAI: number analyzed (Participants) | 1
  UCAI | 0 (0)

11. Secondary Outcome: Rates of Health Care Utilization After Bezlotuxumab Infusion 90 Days
Description: Rates of ED visits and hospital admissions after Bezlotuxumab Infusion 90 Days.
Time Frame: 90 Days
Measure: Number; unit: Ocurrences
Arm/Group | Open Label Bezlotuxumab
Number analyzed (Participants) | 17
Ocurrences
  Hospital admissions | 4
  ED visits | 10

12. Secondary Outcome: Rates of Health Care Utilization After Bezlotuxumab Infusion 12 Months
Description: Rates of ED visits and hospital admissions after Bezlotuxumab Infusion 12 months
Time Frame: 12 months
Measure: Number; unit: Ocurrences
Arm/Group | Open Label Bezlotuxumab
Number analyzed (Participants) | 8
Ocurrences
  ED visits | 6
  Hospital admissions | 2

13. Secondary Outcome: Rates of Health Care Utilization After Bezlotuxumab Infusion 24 Months
Description: Rates of ED visits and hospital admissions after Bezlotuxumab Infusion 24 months
Time Frame: 24 months
Measure: Number; unit: Ocurrences
Arm/Group | Open Label Bezlotuxumab
Number analyzed (Participants) | 5
Ocurrences
  ED visits | 1
  Hospital admissions | 2

ADVERSE EVENTS:
Time Frame: AE data was collected through study completion, an average of 54 weeks.
Arm/Group | Open Label Bezlotuxumab
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT04626947/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT04626947/ICF_001.pdf